CLINICAL TRIAL: NCT01003717
Title: REWARDS-EMI (Registry Experience at the Washington Hospital Center, DES - Endeavor for Myocardial Infarction)
Brief Title: Registry Experience at the Washington Hospital Center, DES - Endeavor for Myocardial Infarction
Acronym: REWARDS-EMI
Status: Completed | Type: Observational
Sponsor: Rebecca Torguson (Other)
Responsible Party: Sponsor-Investigator, Rebecca Torguson, Director, ACRO, Medstar Health Research Institute
Organization: Medstar Health Research Institute (Other)
Other Study IDs: REWARDS EMI
Record Dates: First submitted 2009-10-20; First posted 2009-10-29 (Estimated); Last update posted 2020-01-02 (Actual); Status verified 2019-12

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Endeavor: Patients treated with at least 1 Endeavor, zotarolimus-eluting, Stent as the primary treatment for acute coronary syndrome

SUMMARY:
Single-center registry of patients treated with at least one Endeavor, zotarolimus-eluting, Stent as the primary treatment for acute coronary syndrome at the Washington Hospital Center, with the aim of assessing clinical success and safety at 30 days, 6 months and annually for up to 3 years post Endeavor Stent implantation.

DETAILED DESCRIPTION:
Interventional cardiology was revolutionized by the invention of stents, initially with the bare-metal stents (BMS) and recently with the drug-eluting stents (DES).Zotarolimus-eluting stents have shown promising results in randomized clinical trails, demonstrating a reduction of clinical and angiographic restenosis in comparison to BMS, and comparable clinically-driven target lesion revascularization rates in comparison with Sirolimus-eluting stents. While short-term and 1 year registry data is available from outside of the United States, it will be important to collect "real-world" data regarding the stent usage and outcomes in the United States. In this study we propose to follow patients who received at least one Endeavor® Stent as primary treatment for ACS for up to 3 years post initial stent implantation.

ELIGIBILITY:
Inclusion Criteria:

* Patients, male or female, >18 years of age
* Patients presenting with acute coronary syndrome (ACS), where ACS is defined as ST segment deviation of >1mm or an elevation of the isoenzymes greater than 2x upper limit of normal
* Patients who received at least one Endeavor drug-eluting stent at the Washington Hospital Center

Exclusion Criteria:

* N/A

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who receive at least one Endeavor, zotarolimus-eluting, Stent as the primary treatment for acute coronary syndrome, at the Washington Hospital Center.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2009-10; Primary Completion 2011-10 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
Evaluation of Major Adverse Cardiac Events following implantation of at least one Endeavor, zotarolimus-eluting, Stent as the primary treatment for acute coronary syndrome | Follow Up

CONTACTS AND LOCATIONS:
Overall Officials: Ron Waksman, MD, Principal Investigator — Medstar Research Institute/Cardiovascular Research Institute
Locations (1):
- Washington Hospital Center, Washington D.C., District of Columbia, United States